CLINICAL TRIAL: NCT05924750
Title: A Phase I Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of BL-M11D1 in Relapsed/Refractory Acute Myeloid Leukemia (AML) Patients
Brief Title: A Study of BL-M11D1 in Patients With Relapsed/Refractory Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL-M11D1-101
Record Dates: First submitted 2023-06-16; First posted 2023-06-29 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Relapsed/Refractory Acute Myeloid Leukemia (R/R AML)
MeSH Terms: conditions — Recurrence; Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study treatment (Experimental): Participants receive BL-M11D1 as intravenous infusion for the first cycle (4 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: BL-M11D1

INTERVENTIONS:
Drug: BL-M11D1 — Administration by intravenous infusion

SUMMARY:
Ia: To observe the safety and tolerability of BL-M11D1 in patients with relapsed/refractory acute myeloid leukemia to determine the maximum tolerated dose (MTD) and dose-limiting toxicity (DLT) of BL-M11D1. Ib: Further observe the safety and tolerability of BL-M11D1 at the recommended dose in phase Ia to determine the recommended dose in phase II clinical study (RP2D).

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form and comply with the protocol requirements;
2. No gender restrictions;
3. Age: ≥18 years and ≤75 years;
4. Expected survival time ≥3 months;
5. Histologically and/or cytologically confirmed CD33-positive relapsed/refractory acute myeloid leukemia (AML);
6. Morphological assessment showing ≥5% blasts in the bone marrow;
7. ECOG performance status score ≤2;
8. Peripheral blood white blood cell count ≤25×10^9/L before the first dose;
9. Toxicity from prior anti-tumor therapy has recovered to ≤ Grade 1 as defined by NCI-CTCAE v5.0;
10. Organ function levels meet the requirements within 7 days before the first dose;
11. For premenopausal women with childbearing potential, a pregnancy test (serum/urine) must be performed within 7 days before starting treatment, and the result must be negative; they must not be breastfeeding. All enrolled patients (regardless of gender) must use adequate barrier contraception throughout the treatment period and for 6 months after treatment ends.

Exclusion Criteria:

1. Acute promyelocytic leukemia, acute transformation of chronic myeloid leukemia.
2. Antineoplastic therapy, including chemotherapy, biologic therapy, immunotherapy, definitive radiotherapy, major surgery (investigator-defined), or targeted therapy (including small-molecule tyrosine kinase inhibitors), has been administered within 4 weeks or 5 half-life cycles (whichever is shorter) before the first dose; Or palliative radiotherapy within 2 weeks before the first dose.
3. History of severe heart disease, such as left ventricular ejection fraction < 50%, history of symptomatic congestive heart failure (CHF) ≥ grade 2 (CTCAE v5.0), New York Heart Association (NYHA) ≥ grade 2 heart failure, history of myocardial infarction, unstable angina, etc.
4. Prolonged QT interval (QTc > 450 msec in men or QTc > 470 msec in women), complete left bundle branch block, and III degree atrioventricular block.
5. Active autoimmune diseases and inflammatory diseases, such as systemic lupus erythematosus, psoriasis requiring systemic treatment, rheumatoid arthritis, inflammatory intestinal diseases and Hashimoto's thyroiditis, etc., excluding type I diabetes mellitus, hypothyroidism that can only be controlled by replacement therapy, and skin diseases without systemic treatment (such as vitiligo and psoriasis).
6. Other malignancies diagnosed within 5 years before the first dose, except for radical basal cell carcinoma, squamous cell carcinoma, and/or radical resection carcinoma in situ.
7. Poorly controlled hypertension (systolic blood pressure > 150 mmHg or diastolic blood pressure > 100 mmHg).
8. Patients with pulmonary disease grade ≥3 defined by CTCAE v5.0, current or previous interstitial lung disease (ILD).
9. Patients with central nervous system involvement.
10. Patients with a history of allergy to recombinant humanized antibody or human-mouse chimeric antibody or to any of the ingredients of BL-M11D1.
11. Prior organ transplantation or allogeneic hematopoietic stem cell transplantation (Allo-HSCT).
12. Human immunodeficiency virus (HIVAb) positive, active tuberculosis, active hepatitis B virus infection (HBsAg positive; HBcAb positive and HBV-DNA copy number > lower detection limit) or active hepatitis C virus infection (HCV antibody positive and HCV-RNA > lower detection limit).
13. Active infection requiring systemic treatment, such as severe pneumonia, bacteremia, sepsis, etc.
14. Presence of pleural, abdominal, pelvic or pericardial effusion with clinical symptoms or requiring repeated drainage.
15. Had participated in another clinical trial within 4 weeks before the first dose (calculated from the time of last dose).
16. Pregnant or lactating women.
17. Other conditions for participation in the trial were not considered appropriate by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2023-08-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Phase Ia: Dose limiting toxicity (DLT) | Up to 28 days after the first dose
  DLTs are assessed according to NCI-CTCAE v5.0 during the first cycle and defined as occurrence of any of the toxicities in DLT definition if judged by the investigator to be possibly, probably or definitely related to study drug administration.
Phase Ia: Maximum tolerated dose (MTD) | Up to 28 days after the first dose
  MTD is defined as the highest dose level at which no more than 1 in 6 participants experienced a DLT during the first cycle .
Phase Ib: Recommended Phase II Dose (RP2D) | Up to 28 days after the first dose
  The RP2D is defined as the dose level chosen by the sponsor (in consultation with the investigators) for phase II study, based on safety, tolerability, efficacy, PK, and PD data collected during the dose escalation study of BL-M11D1.

SECONDARY OUTCOMES:
Treatment-Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of BL-M11D1. The type, frequency and severity of TEAE will be evaluated during the treatment of BL-M11D1.
Cmax | Up to 28 days after the first dose
  Maximum serum concentration (Cmax) of BL-M11D1 will be investigated.
Tmax | Up to 28 days after the first dose
  Time to maximum serum concentration (Tmax) of BL-M11D1 will be investigated.
T1/2 | Up to 28 days after the first dose
  Half-life (T1/2) of BL-M11D1 will be investigated.
AUC0-t | Up to 28 days after the first dose
  AUC0-t is defined as area under the serum concentration-time curve from time 0 to the time of the last measurable concentration.
CL (Clearance) | Up to 28 days after the first dose
  CL in the serum of BL-M11D1 per unit of time will be investigated.
Ctrough | Up to 28 days after the first dose
  Ctough is defined as the lowest serum concentration of BL-M11D1 prior to the next dose will be administered.
ADA (anti-drug antibody) | Up to approximately 24 months
  ADA of BL-M11D1 will be evaluated.
Phase Ib: Objective Response Rate (ORR) | Up to approximately 24 months
  ORR is defined as the percentage of participants, who has a CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experiences a confirmed CR or PR is according to RECIST 1.1.
Phase Ib: Disease Control Rate (DCR) | Up to approximately 24 months
  The DCR is defined as the percentage of participants who has a CR, PR, or Stable Disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD]).
Phase Ib: Duration of Response (DOR) | Up to approximately 24 months
  The DOR for a responder is defined as the time from the participant's initial objective response to the first date of either disease progression or death, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Junyuan Qi, PHD, Principal Investigator — Institute of Hematology and Blood Diseases Hospital, Chinese Academy of Medical Sciences; Jianxiang Wang, MS, Principal Investigator — Institute of Hematology and Blood Diseases Hospital, Chinese Academy of Medical Sciences
Locations (8):
- China (8):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Beijing Hospital, Beijing, Beijing Municipality
  - Institute of Hematology, the First Hospital of Harbin, Haerbin, Heilongjiang
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shangdong
  - Shanghai Tongji Hospital, Shanghai, Shanghai Municipality
  - West China Hospital，Sichuan University, Chengdu, Sichuan
  - Institute of Hematology and Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality